CLINICAL TRIAL: NCT04094558
Title: Validation of the Small Intestine Microbiome Aspiration (SIMBA) Capsule
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Nimble Science Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 19-0957
Record Dates: First submitted 2019-09-17; First posted 2019-09-19 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-06

CONDITIONS: Proof of Concept; Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IBS-D (Active Comparator): Participant diagnosed with Irritable Bowel Syndrome, diarrhea predominant, confirmed by study doctors using Rome IV criteria.
  Interventions: Device: Ingestible capsule; Procedure: Sedated EGD; Diagnostic Test: Lactulose Breath Test
- IBS-C (Active Comparator): Participant diagnosed with Irritable Bowel Syndrome, constipation predominant, confirmed by study doctors using Rome IV criteria.
  Interventions: Device: Ingestible capsule; Procedure: Sedated EGD; Diagnostic Test: Lactulose Breath Test
- Healthy Control (Active Comparator): Participant with no ongoing medical conditions affecting GI health.
  Interventions: Device: Ingestible capsule; Procedure: Sedated EGD; Diagnostic Test: Lactulose Breath Test

INTERVENTIONS:
Device: Ingestible capsule — Participants will swallow capsules and collect in stool concurrent with stool samples
Procedure: Sedated EGD — Participants will undergo sedated esophagogastroduodenoscopy (EGD) for collection of small intestine aspirate and simultaneous saliva sample.
Diagnostic Test: Lactulose Breath Test — Hydrogen and methane breath test with lactulose substrate

SUMMARY:
Prospective, open label trial to establish the ability of the SIMBA Capsule to accurately obtain a sample from the small bowel of participants with IBS (10 constipation-predominant (IBS-C) and 10 diarrhea-predominant (IBS-D)) and healthy participants (n=10). The accuracy of targeting the small bowel will be established by visual confirmation via X-ray. The clinical utility of the collected sample will be evaluated by analysis with samples obtained by the current gold standard (duodenal aspirate), as well as stool analysis and LBT.

ELIGIBILITY:
Inclusion Criteria

1. Aged between 18 and 70 years.
2. Diagnosis of IBS by Rome 4 criteria (IBS groups) or no previous diagnosis of IBS or suspected IBS (Control group).
3. Ability to understand and provide informed consent.
4. Ability and willingness to meet the required schedule and study interventions.
5. No planned change in diet or medical interventions during the study duration.
6. Adequate mobility to transfer repeatedly between X-ray (standing or lying), and waiting (sitting).
7. Willing and able to undergo a sedated esophagogastroduodenoscopy (EGD) with aspirate and brushing.

Exclusion Criteria

1. Prior gastrointestinal disease, surgery, or radiation treatment which, in the investigator's opinion, would lead to intestinal structuring or obstruction with a risk of capsule non-excretion (particular diseases which would be assessed on a case-by-case basis would include, achalasia, eosinophilic esophagitis, Crohn's disease, cancer diagnosis or treatment within the past year, or previous esophageal, gastric, small intestinal, or colonic surgery. Appendectomy or cholecystectomy more than 3 months prior to enrollment are acceptable).
2. Use of any medications in the previous week that could substantially alter gastrointestinal motor function (e.g., opioids, prokinetics, anticholinergics, laxatives), or acidity (PPI, H2RA).
3. History of oropharyngeal dysphagia or other swallowing disorder with a risk of aspiration of the capsule.
4. Females of childbearing age who are not practicing birth control and/or are pregnant or lactating.
5. No antibiotics, or colon cleanses/bowel prep for 2 weeks.
6. < 2 bowel movements per week (Control Group).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-10-27 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2022-06-16 (Actual)

PRIMARY OUTCOMES:
Bacterial composition | same day
  1. Correlations of bacterial composition (superimposability of PLS-DA mapping) of samples collected by the SIMBA Capsule compared to small bowel aspirate and to mucosal microbiome sample obtained by brushing. (hypothesis: findings will be similar)
Bacterial composition | same day
  2. Correlations of bacterial composition (superimposability of PLS-DA mapping) of samples collected by the SIMBA Capsule compared to stool sample obtained at same time. (hypothesis: findings will be different)

SECONDARY OUTCOMES:
Bacterial composition | within 5 days of primary measures
  1. Correlation of hydrogen- and methane-producing bacteria species (by 16s RNA sequencing) found by SIMBA Capsule with hydrogen and methane concentrations (peak and rise in ppm) detected by LBT and bacterial density (CFU/ml) of endoscopic aspirate.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher N Andrews, Principal Investigator — Cumming School of Medicine, University of Calgary
Locations (1):
- Cumming School of Medicine, University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No